CLINICAL TRIAL: NCT06457815
Title: Iron Deficiency in Acute Myocardial Infarction: Prevalence Pilot Study
Acronym: IDAMI Pilot
Status: Recruiting | Type: Observational
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ACU020
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myocardial Infarction - Type 1: Patients presenting with acute MI will have a blood test to understand their iron status.

SUMMARY:
Acute Myocardial Infarction (heart attacks) affect about 86000 people each year in the UK. Given this large number of people, it is important that health teams look at ways to ensure the best care to improve outcomes after a heart attack.

In related heart conditions, the role of iron is important, but there isn't much information about what effect iron levels have on patients following a heart attack.

We want to plan a large scale study to look at this, but need some early data to understand how many patients have low iron levels. This small study will take part at one NHS Trust and will test for iron levels in all patients who provide consent (we expect up to 70 patients will take part). We will also collect data from medical notes for these patients and use all of this information together to understand more about iron and to plan a larger study.

ELIGIBILITY:
Inclusion:

1. - Adults patients who sign an informed consent form.
2. - Type 1 myocardial infarction within the previous 10 days

Exclusion

1 - Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of iron deficiency | within 10 days of acute MI
  Prevalence of iron deficiency in a population of patients following acute MI.

CONTACTS AND LOCATIONS:
Overall Officials: David Austin, MD, Principal Investigator — South Tees Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, Teesside
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: Undecided